CLINICAL TRIAL: NCT07031245
Title: Reducing Burnout Among VA PCPs Using Evidence-Based Quality Improvement
Brief Title: Evidence-Based Quality Improvement to Reduce VA Primary Care Burnout
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Eric A. Apaydin, Research Health Scientist, VA Greater Los Angeles Healthcare System
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: CDA 21-158; IK2HX003534 (NIH)
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-07

CONDITIONS: Burnout; Burnout Syndrome
Keywords: primary care; VA; burnout; EBQI; evidence-based; quality improvement
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Four-year modified stepped wedge trial with three interventions sites, separated by one year, and two control sites across the four years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evidence-based quality improvement (EBQI) (Experimental): Evidence-based quality improvement (EBQI) to facilitate the development and implementation of one or more burnout reduction interventions. The EBQI-facilitated interventions will be actively managed my the research team for one year, and may be passively continue by clinic leadership, providers, and staff for the following years.
  Interventions: Behavioral: Evidence-based quality improvement (EBQI)
- Usual care (No Intervention): Researchers will have no interaction with the clinics beyond survey administration.

INTERVENTIONS:
Behavioral: Evidence-based quality improvement (EBQI) — Evidence-based quality improvement (EBQI) is a multi-level implementation strategy that aids in the development and implementation of evidence-based interventions to reduce burnout. Preliminary survey, interview, and systematic review data on burnout, turnover intent, burnout drivers, and burnout interventions will be presented to an expert panel for each intervention site. These panels will collectively decide on the top categories of burnout drivers to target and burnout interventions to implement. These top drivers and intervention categories will be presented to site-level providers and staff and proposals will be solicited for quality improvement (QI) interventions to reduce burnout that reflect these categories and address these drivers. The expert panels will then choose one or more of these QI interventions to implement and evaluate at each intervention site.
  Arms: Evidence-based quality improvement (EBQI)

SUMMARY:
Burnout is highly prevalent among VA primary care providers and staff, impairing productivity and retention, as well as safety, quality, and patient experience. In this pilot trial, the investigators will facilitate the development of burnout reduction interventions using an evidence-based quality improvement (EBQI) approach, and then evaluate the feasibility, acceptability and effectiveness of a pilot EBQI-facilitated burnout reduction intervention in a modified stepped wedge design in one VA region.

DETAILED DESCRIPTION:
Burnout, a long-term psychological response to chronic workplace stress, is highly prevalent among providers and staff in VA primary care. Healthcare worker (HCW) burnout is not only detrimental to affected individuals, but also to the organizations that they work in. High rates of HCW burnout are linked to increased medical errors, worse quality of care, and worse patient experience. Burned out HCWs also work fewer hours and are more likely to leave their organization. Organizational interventions to reduce burnout are more effective than individual interventions, but no single organizational intervention is applicable to all settings. The investigators propose to use evidence-based quality improvement (EBQI) to utilize collaborative leadership and PACT teamlet input to develop and pilot test a burnout reduction intervention, informed by evidence and facilitated by experts, that is tailored to the specific needs of participating primary care clinics. Findings from this work will inform strategies for implementing burnout interventions in other VA facilities, adapted to local organizational contexts.

In VA, 31-55% of providers, nurses, clinical associates, and administrative associates in patient-aligned care team (PACT) teamlets consistently report burnout. Strong primary care models are essential to the VA's integrated delivery system. High burnout, and subsequent turnover, could erode that strength by decreasing primary care staffing, team function and PACT fidelity, thereby impairing Veteran access and shifting more care to the community. Addressing burnout in primary care before it leads to larger downstream effects is essential to preserving Veteran health and the integrity of the VA healthcare system. In addition, addressing burnout in primary care meets the HSR&D and ORD research priorities of primary care practice and complex chronic disease management, and of increasing substantial real-world impact of VA research. Innovation: EBQI is an effective and well-evaluated strategy that aided in the implementation of PACT, Women's Health PACT, depression collaborative care, and smoking cessation guidelines. The strategy also reduced provider and staff burnout during PACT implementation, but has never been used in tandem with burnout interventions to optimize impacts. This project is the first endeavor to combine EBQI as an implementation strategy with evidence-based burnout interventions, adapted for local organizational contexts. Through EBQI, a multi-level, collaborative approach that empowers frontline HCWs, the investigators may increase the feasibility and impact of burnout reduction interventions.

The investigators will conduct a pilot, modified stepped wedge trial of EBQI for primary care burnout in 5 primary care clinics (based in 2 VA Medical Centers and 3 community-based outpatient clinics) in 2 VA healthcare systems in 1 Veterans Integrated Service Network. Three intervention sites will implement EBQI-facilitated interventions to reduce burnout, while 2 control sites will receive usual care. Survey data on burnout, drivers of burnout, turnover intent, intervention feasibility and acceptability, and other survey respondent individual and workplace characteristics will be collected annually through the trial period.

ELIGIBILITY:
Site Inclusion Criteria:

* 5 primary care clinics (2 VA Medical Centers [VAMCs] and 3 community-based outpatient clinics [CBOCs]) in 2 VA healthcare systems in 1 VA Veterans Integrated Service Network

Provider and Staff Inclusion Criteria:

* Primary care providers, registered nurses, clinical associates (e.g., licensed vocational or practical nurses), or administrative associates (e.g., clerks) on regular Patient-Aligned Care Team (PACT) teamlets at a study site.

Site Exclusion Criteria:

* All other VAMCs and CBOCs.

Provider and Staff Exclusion Criteria:

* Other primary care professionals at a study site.
* Members of special types of PACT teamlets at a study site.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 203 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Burnout | Annually, from enrollment until the end of the study, three years later (4 survey administrations).
  22-item Maslach Burnout Inventory.
  Minimum score of 0 for all domains. Maximum score of 54 for emotional exhaustion domain. Maximum score of 30 for depersonalization domain. Maximum score of 48 for personal accomplishment domain.
  Higher scores are worse, except for the personal accomplishment domain where higher scores are better.

SECONDARY OUTCOMES:
Turnover intent | Annually, from enrollment until the end of the study, three years later (4 survey administrations).
  Turnover intent in the next year, and factors related to turnover intent (questions adapted from the VA All Employee Survey).
Workplace drivers of burnout | Annually, from enrollment until the end of the study, three years later (4 survey administrations)
  28-item Areas of Worklife Survey. Minimum score of 0 for all domains. Maximum score of 25 for workload domain. Maximum score of 20 for control domain. Maximum score of 20 for reward domain. Maximum score of 25 for community domain. Maximum score of 30 for fairness domain. Maximum score of 20 for values domain. Higher scores are better for all domains.
Depression | Annually, from enrollment until the end of the study, three years later (4 survey administrations)
  14-item Hospital Anxiety and Depression Scale. Minimum score of 0 for depression domain. Maximum score of 21 for depression domain. Higher scores are worse.
Anxiety | Annually, from enrollment until the end of the study, three years later (4 survey administrations)
  14-item Hospital Anxiety and Depression Scale. Minimum score of 0 for anxiety domain. Maximum score of 21 for anxiety domain. Higher scores are worse.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Bakersfield VA Clinic, VA Greater Los Angeles Healthcare System, Bakersfield, California
  - Tibor Rubin VA Medical Center, VA Long Beach Healthcare System, Long Beach, California
  - West Los Angeles VA Medical Center, VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Sepulveda VA Medical Center, VA Greater Los Angeles Healthcare System, North Hills, California
  - Santa Maria VA Clinic, VA Greater Los Angeles Healthcare System, Santa Maria, California

IPD SHARING:
Plan to Share IPD: No
Study data is confidential and cannot be shared outside of the VA.